CLINICAL TRIAL: NCT06662799
Title: Intraoperative Reduction of Ventilation of Dorsal Lung Regions and Postoperative Pulmonary Complications After Laparoscopic Colorectal Cancer Surgery
Brief Title: Dorsal Vetilation and PPCs in Colorectal Cancer Surgery Patients
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, xiangming fang, Director of the Anesthesiology Department, First Affiliated Hospital of Zhejiang University
Other Study IDs: IIT20240443B
Record Dates: First submitted 2024-10-07; First posted 2024-10-29 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Surgery; Postoperative Pulmonary Complications (PPCs)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Postoperative pulmonary complications (PPCs) are common in patients after major abdominal surgery. It has been shown that 5-40% of patients occur PPCs after major surgery, and the mid to high PPC rate is observed after laparoscopic colorectal cancer surgery. PPCs are associated with poor clinical outcomes including prolonged hospital length of stay and increased morbidity and mortality.

Mechanical ventilation during general anesthesia can lead to a redistribution of ventilation, increase the aereation in the ventral parts of the lung, whereas reduce ventilation in the dorsal parts of the lung compared with spontaneous breathing (SB) in the awake state in supine position. The reduction of ventilation of dorsal lung regions indicates the presence of dorsal atelectasis during mechanical ventilation after general anesthesia, which may be associated with PPCs. However, there is still no evidence to reveal the association between the reduction of dorsal ventilation and PPCs.

Recently, electrical impedance tomography (EIT), which allows visualization of lung ventilation in real time, and assessment of regional lung ventilation. It is feasible to assess the change of ventral/dorsal lung ventilation during the surgery using EIT. To date, no study has investigated whether the change of ventral/dorsal lung ventilation revealed by EIT could be associated with PPCs.

So, this prospective observational study aims to clarify whether patients developing postoperative pulmonary complications had higher reduction of dorsal lung ventilation during operation after general anesthesia as compared to patients not developing postoperative pulmonary complications. Ratio of dorsal ventilation during spontaneous respiration (T0) in the awake state as a reference, the proportion of dorsal ventilation after anesthesia induction and endotracheal intubation (T1), body position change and capnoperitoneum (T2), and at the end of surgery (T3) were analyzed. Thereafter, evaluating the change of dorsal ventilation in patients with PPCs and without PPCs at different time points.

According to the method of sample size calculation published by Scaramuzzo G et al. (Anesthesiology. 2024 Oct 1;141(4):693-706.). A minimum sample size required for this study was calculated as following: using the difference of reduction of dorsal ventilation at the end of surgery between the patients with PPCs and non-PPCs as the primary outcome. Considering the data of our preliminary experiment showed that a reduction of dorsal lung ventilation at the end of surgery is 12 ± 6% and hypothesizing 30% of patients experiencing postoperative pulmonary complications and a relative clinically relevant increase in reduction of dorsal lung ventilation of 40% in those with postoperative pulmonary complications, we found that 83 patients were sufficient to evaluate differences between groups (effect size 0.8) with a power of 0.90 and an α error of 0.05. Considering a dropout of 10%, we found a minimum sample size of 92 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* ASA grade I-III
* The patients who are planning to undergo laparoscopic colorectal cancer surgery

Exclusion Criteria:

* Emergency surgery
* Time of surgery less than 2 hours
* Preoperatively present upper respiratory tract infection or acute pulmonary infection
* Previous history of pulmonary surgery
* Preoperative use of home ventilator
* Inability to perform EIT monitoring
* Declined to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing laparoscopic colorectal cancer surgery
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
The difference of reduction of dorsal ventilation at the end of surgery between the patients with PPCs and non-PPCs | 1-7 days after surgery.
  1. EIT to monitor the regional ventilation of the patients at spontaneous breathing (SB) in the awake state in supine position (T0) and the end of surgery (T3). The reduction of the ratio of dorsal ventilation will be caculated between T3 and T0.
  2. Follow-up the patients untill discharge from the hostiptal. Based on whether pulmonary complication occurs during 7 days after surgery, the participants will be divided into the patients with PPCs and the patients with non-PPCs.
  3. The difference of reduction of dorsal ventilation at the end of surgery (T3) between the patients with PPCs and non-PPCs will be analyzed.

SECONDARY OUTCOMES:
The difference of reduction of dorsal ventilation at endotracheal intubation after general anesthesia induction between the patients with PPCs and non-PPCs | 1-7 days after surgery.
  EIT to monitor the regional ventilation of the patients at spontaneous breathing (SB) in the awake state in supine position (T0) and endotracheal intubation after general anesthesia induction (T1). The reduction of the ratio of dorsal ventilation will be caculated between T1 and T0. 2. Follow-up the patients untill discharge from the hostiptal. Based on whether pulmonary complication occurs during 7 days after surgery, the participants will be divided into the patients with PPCs and the patients with non-PPCs. 3. The difference of reduction of dorsal ventilation at endotracheal intubation after general anesthesia induction (T1) between the patients with PPCs and non-PPCs will be analyzed.
The difference of reduction of dorsal ventilation at pneumoperitoneum and body position change between the patients with PPCs and non-PPCs | 1-7 days after surgery.
  EIT to monitor the regional ventilation of the patients at spontaneous breathing (SB) in the awake state in supine position (T0) and pneumoperitoneum and body position change (T2). The reduction of the ratio of dorsal ventilation will be caculated between T2 and T0. 2. Follow-up the patients untill discharge from the hostiptal. Based on whether pulmonary complication occurs during 7 days after surgery, the participants will be divided into the patients with PPCs and the patients with non-PPCs. 3. The difference of reduction of dorsal ventilation at pneumoperitoneum and body position change (T2) between the patients with PPCs and non-PPCs will be analyzed.
The risk factors which are associated with PPCs | 1-7 days after surgery.
  1. Collecting age, gender, height, weight, history of chronic diseases such as hypertension and chronic obstructive pulmonary disease (COPD) etal, and assessing the pre-operative respiratory risk of patients using the ARISCAT (Assess Respiratory Risk in Surgical Patients in Catalonia) scoring system developed by Canet J et al.
  2. To explore the independent risk factors which are associated with PPCs using logistic regression.

OTHER OUTCOMES:
The difference of hostpital stays between the patients with PPCs and non-PPC | From the end of surgery to the discharge from hospital, an average of 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The first Affiliated Hospital, School of Medicine, Zhejiang University., Hangzhou, Zhejiang, China